CLINICAL TRIAL: NCT05056805
Title: "SurgeryStrong". Preoperative Strength Exercise and Nutrition Program in Patients Completing Neoadjuvant Chemoradiation Therapy for Pancreatic and Gastric Cancer: A Randomized Trial Testing Effects on Strength, Fitness, Health-Related Quality of Life, and Perioperative Outcomes
Brief Title: An Exercise and Nutrition Monitoring Intervention (Pt Pal) for the Improvement of Strength in Patients With Pancreatic or Stomach Cancer Receiving Chemoradiation Therapy Before Surgery, SurgeryStrong Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0026; NCI-2021-02655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0026 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2022-10

CONDITIONS: Gastric Adenocarcinoma; Pancreatic Adenocarcinoma
MeSH Terms: interventions — Exercise; Diet Therapy; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (aerobic exercise, nutritional recommendation) (Active Comparator): Patients are encouraged to complete at least 30 minutes of moderate intensity aerobic exercise, at least 3 times per week. Patients receive nutrition consultation with a registered dietitian and monitor dietary intake. Aerobic exercises and nutrition are tracked in the Pt Pal app
  Interventions: Other: Aerobic Exercise; Other: Nutritional Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (aerobic, strength exercise, nutritional recommendation) (Experimental): Patients complete at least 30 minutes of moderate intensity aerobic exercise (such as brisk walking or stationary bike cycling) at least 3 times per week. Patients also complete strength exercises with resistance tubes/bands at least 2 times per week, with at least 2 sets of 8-15 repetitions of the exercises taught. Patients receive nutrition consultation with a registered dietitian and monitor dietary intake. Patients also consume a high protein snack/meal/shake (15-25 grams) within 1 hour after any strengthening exercises. Exercise activities and nutrition are tracked in the Pt Pal app.
  Interventions: Other: Aerobic Exercise; Other: Dietary Intervention; Other: Nutritional Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Aerobic Exercise — Receive aerobic exercise encouragement
  Other Names: Aerobic Activity
Other: Dietary Intervention — Consume high protein snack/meal/shake
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm B (aerobic, strength exercise, nutritional recommendation)
Other: Nutritional Intervention — Receive nutritional consultation and guidelines
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Complete strengthening exercise
  Other Names: Strength Training
  Arms: Arm B (aerobic, strength exercise, nutritional recommendation)

SUMMARY:
This clinical trial studies the effectiveness of a home-based exercise and nutrition monitoring program called Pt Pal in improving strength in patients with pancreatic or stomach cancer receiving chemoradiation therapy before surgery. Pt Pal is a mobile health technology used to facilitate communication between the care team and the patient/caregiver, by allowing the care team to send from their web-portal, exercise routines, activities of daily living, diet recommendations, surveys and educational material to the patient/caregiver's mobile device. The Pt Pal application (app) then captures the patient/caregiver activity adherence data and reports those results back to the care team. The Pt Pal program may help improve overall strength in patients undergoing surgery for pancreatic and stomach cancer relative to standard care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. In patients with pancreatic and gastric cancer undergoing preoperative chemoradiation and potentially curative resection, compare the change in dynamic lower muscle strength as measured by the 1 repetition maximum (1-RM) leg press between the time of enrollment and prior to resection in those who: a. Are offered aerobic exercise encouragement prior to surgery b. Are offered aerobic exercise encouragement, nutrition monitoring, and a structured strength exercise program prior to surgery.

SECONDARY OBJECTIVES:

I. To compare the change in dynamic muscle strength as measured by the 1-RM for the chest press, seated row, and leg extension.

II. To compare upper and lower body muscle endurance as defined by the maximal number of repetitions performed at 70% of the pre-exercise 1-RM for the chest and leg press.

III. To compare the change in the six minute walk test (6MWT) distance of patients between the time of enrollment and prior to resection.

IV. To compare physical function (patient-reported based on the Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form and objectively based on grip strength) between groups.

V. To compare the quality of life (Functional Assessment of Cancer Therapy, patients with hepatobiliary cancer [FACT-Hep]) between groups.

VI. To compare exercise motivation (Behavioral Regulation in Exercise Questionnaire [BREQ]-3) between groups.

VII. To compare anthropometric measures (e.g., weight, skeletal muscle, visceral fat and subcutaneous fat) using SliceOMatic software from usual care computed tomography (CT) scans between groups.

VIII. To assess the incidence of perioperative adverse events that occur within 90 days between groups (Accordion score).

IX. To compare changes in physical activity between the time of enrollment and immediately prior to surgery based on the Modified Godin-Shephard Leisure Time Physical Activity Questionnaire.

X. To evaluate feasibility of patient completion of 24-hour recall via Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA-24).

XI. To measure adoption of nutrition recommendations as compared to baseline. XII. To compare adherence to nutrition recommendations within and between groups.

XIII. To compare "usual care" laboratory studies including those that are indicators of nutritional status within and between groups.

XIV. To compare the vascular and tumor structure, and immune cell infiltration in tumors between patients in different groups.

XV. To compare potential biomarkers of angiogenesis and inflammation that correlate with exercise, disease pathology, and/or clinical and functional outcomes.

XVI. To store in a research bank any remaining tissue or blood (collected for the purposes of the above objectives) for the possibility of future analysis.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients are encouraged to complete at least 30 minutes of moderate intensity aerobic exercise, at least 3 times per week. Patients receive nutrition consultation with a registered dietitian and monitor dietary intake. Aerobic exercises and nutrition are tracked in the Pt Pal app.

ARM B: Patients complete at least 30 minutes of moderate intensity aerobic exercise (such as brisk walking or stationary bike cycling) at least 3 times per week. Patients also complete strength exercises with resistance tubes/bands at least 2 times per week, with at least 2 sets of 8-15 repetitions of the exercises taught. Patients receive nutrition consultation with a registered dietitian and monitor dietary intake. Patients also consume a high protein snack/meal/shake (15-25 grams) within 1 hour after any strengthening exercises. Exercise activities and nutrition are tracked in the Pt Pal app.

After randomization, patients are followed up at 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic or gastric adenocarcinoma, biopsy-proven
* Have completed or are within 2 weeks of completion of preoperative chemoradiotherapy either on- or off-protocol
* Anticipated to undergo potentially curative resection in 4-6 weeks from enrollment
* Able to understand the description of the study and willing to participate
* Able to understand the exercise program
* Able to independently maintain daily exercise logs via Pt Pal -iOS, Android or desktop web browser on their own personal device
* Telephone or email access and agreement to engage with the research personnel via phone or email
* Meet all screening requirements, including physician clearance
* >= age 18

Exclusion Criteria:

* Non-English speaking
* Has participated in moderate to high intensity strengthening exercises at least two times per week within the past four weeks prior to enrollment
* Unable to complete the baseline assessment questionnaires or functional assessments
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV)
* Recent fracture or acute musculoskeletal injury that precludes the ability to weight bear fully on all 4 limbs in order to participate in an exercise intervention
* Numeric pain rating scale of >= 7 out of 10
* Myopathic or rheumatologic disease that impacts physical function
* Recurrent cancer following prior resection
* < age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Change in dynamic lower muscle strength | through study completion, an average of a year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H Katz, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT05056805/ICF_000.pdf